CLINICAL TRIAL: NCT06020885
Title: Fraction Dose Escalation of Split-course Hypofractionated Concurrent Chemoradiotherapy Following Induction Chemo-immunotherapy in Unresectable Locally Advanced Esophageal Squamous Carcinoma: a Phase I Study.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-10102
Record Dates: First submitted 2023-08-26; First posted 2023-09-01 (Actual); Last update posted 2025-07-21 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Split-course hypofractionated concurrent chemoradiotherapy; Fraction dose escalation; Induction chemo-immunotherapy; Unresectable locally advanced esophageal squamous carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experiment group (Experimental): This is a prospective, single-arm, phase 1 trial. A total of 18 unresectable LA-ESCC patients are required to be enrolled.
  1. Induction chemo-immunotherapy All patients receive 2-3 cycles of Abraxane 260mg/m2 d1+cisplatin 60mg/m2 d1+Toripalimab 240mg d1.
  2. Hypo-CCRT Evaluation will be performed three weeks after the induction chemo-immunotherapy, LA-ESCC patients without disease progression will continue the split-course hypo-CCRT treatment.
  Split-course hypo-CCRT is administered at the following three dose levels:
  * Level 1: DT 3000cGy/10 daily fractions/300cGy in the first course, DT 2000cGy/10 daily fractions/200cGy in the second course;
  * Level 2: DT 2800cGy/7 daily fractions/400cGy in the first course, DT 2200cGy/10 daily fractions/220cGy in the second course;
  * Level 3: DT 2500cGy/5 daily fractions/500cGy in the first course, DT 2500cGy10 daily fractions/250cGy in the second course.
  Interventions: Radiation: Split-course hypo-CCRT; Drug: Induction chemo-immunotherapy; Drug: Concurrent chemotherapy

INTERVENTIONS:
Radiation: Split-course hypo-CCRT — Split-course hypo-CCRT is administered at the following three dose levels:
  * Level 1: DT 3000cGy/10 daily fractions/300cGy in the first course, DT 2000cGy/10 daily fractions/200cGy in the second course;
  * Level 2: DT 2800cGy/7 daily fractions/400cGy in the first course, DT 2200cGy/10 daily fractions/220cGy in the second course;
  * Level 3: DT 2500cGy/5 daily fractions/500cGy in the first course, DT 2500cGy10 daily fractions/250cGy in the second course.
Drug: Induction chemo-immunotherapy — All patients receive 2-3 cycles of Abraxane 260mg/m2 d1+cisplatin 60mg/m2 d1+Toripalimab 240mg d1.
Drug: Concurrent chemotherapy — Concurrent capecitabine was administered orally at 1000mg/m2 twice daily within half an hour after meals concurrently with radiotherapy.

SUMMARY:
This Phase I study is to determine the maximum tolerated fraction dose (MTD) for split-course hypo-CCRT following induction chemo-immunotherapy in LA-ESCC patients, to clarify the dosimetric advantage of split-course hypo-CCRT, and to investigate the treatment-related toxicities and quality of life of the new regimen.

DETAILED DESCRIPTION:
This Phase I study is to determine the maximum tolerated fraction dose (MTD) for split-course hypo-CCRT following induction chemo-immunotherapy in LA-ESCC patients, to clarify the dosimetric advantage of split-course hypo-CCRT, and to investigate the treatment-related toxicities and quality of life of the new regimen.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed ESCC
* II-IVB stages (IVB stage only with metastatic celiac or supraclavicular lymph nodes) based on the TNM staging system proposed by the International Union Against Cancer (UICC 2002)
* Eastern Cooperative Oncology Group (ECOG) performance status score 0-1
* Charlson Comorbidity Index score≤4
* oral medication can be administered despite esophageal obstruction
* adequate hematological, renal and hepatic functions

Exclusion Criteria:

* contraindication for radiotherapy or chemotherapy
* prior malignancies, except for curable non-melanoma skin cancer or cervical carcinoma in situ
* distant metastasis, except for celiac or supraclavicular lymph nodes metastases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Tolerated fraction dose | 6 months
  Define the maximum tolerated fraction dose (MTD) for split-course hypo-CCRT following induction chemo-immunotherapy.

SECONDARY OUTCOMES:
2-year overall survival rate | 2-year
2-year progression-free survival rate | 2-year
Clinical response rate | 2 months after radiotherapy
  The percentage of patients who had partial remission or complete remission after therapy
The rate of grade 3 or 4 toxicities according to CTCAE5.0 | 1 year after therapy
  the percentage of patients who develop grade 3 or 4 toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Professor, Principal Investigator — Sun yat-sen universtiy cancer center
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China